CLINICAL TRIAL: NCT03667612
Title: Endogenous Mechanisms of Inactivation of the Endothelium Tumor
Acronym: BreastIls
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Institut de Biologie de Lille (Other)
Responsible Party: Sponsor
Other Study IDs: BreastIls-1605
Record Dates: First submitted 2018-09-05; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer; Colon Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA from tumor samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with breast cancer: * Patients clinical data collection
  * Selection of patients tumor samples and centralization at the Oscar Lambret and the Henri Becquerel centres
  * Realization of tumor samples series of cuts and paraffin shavings for:
    * Quantitative RT-PCR (Reverse Transcription PCR): Assessment of the expression of the genes regulating the endothelium activation: egfl7, SetD5 (SET Domain Containing 5), other genes and microRNAs identified in the high-throughput screen realized by the Dr. F Soncin
    * Semi-quantitative evaluation of the same genes expression by in situ hybridization techniques (if probes available)
    * Semi-quantitative evaluation of the expression of the corresponding proteins by immunohistochemistry techniques (If antibodies available)
    * Characterization of lymphocyte populations
    * Measurement of the endothelial cell density, the lymphatic endothelium and the "High Endothelial Venules"
- Patients with colorectal cancer: * Patients clinical data collection
  * Selection of patients tumor samples and centralization at the Oscar Lambret Center and the Henri Becquerel Center by the teams of Dr. Yves-Marie Robin and Jean-Michel Picquenot, Head of the Anatomy and Cytopathology Departments
  * Realization of series of cuts and paraffin shavings of the tumor samples for:
    * Quantitative RT-PCR: Assessment of the expression of the genes regulating the endothelium activation: egfl7, SetD5, other genes and microRNAs identified in the high-throughput screen realized by the Dr. F Soncin
    * Semi-quantitative evaluation of the same genes expression by in situ hybridization techniques (if probes are available)
    * Semi-quantitative evaluation of the expression of the corresponding proteins by immunohistochemistry techniques (If antibodies are available)
    * Characterization of lymphocyte populations
    * Measurement of the endothelial cell density, the lymphatic endothelium and the "High Endothelial Venules"

SUMMARY:
The role of immunity in the development of cancers, and the associated escape mechanisms, have attracted renewed interest since the publication of tests testing immunological checkpoint inhibitors. One of the steps in the probably least studied immunological response is the penetration of immunocompetent cells within the tumor across the vascular barrier. This infiltration is suggested as a prognostic and predictive marker of treatment response, particularly in triple negative HER2 (Human Epidermal Growth Factor Receptor-2) overexpressing breast cancers. The methods of evaluating these infiltrates are complex and have been the subject of recommendations.

A better understanding of the mechanisms of infiltration of immunity cells within tumors will certainly help to better understand the impact of cancer treatments and develop new therapeutic strategies.

It is this issue of vascular endothelium that Dr. Soncin's team is developing as part of an INCa (Institut National du cancer) project. The egfl7 / VE-statin (vascular endothelial-statin) gene is thought to be involved in transendothelial passage of immune cells from vascular lumen to tumor. Its expression has already been studied in a series of breast cancers. Other markers of endothelial activation are currently being identified.

The main objective of this project will be to better understand the behavior of the endothelium in a population of breast cancer where the infiltrate in immune cells is precisely likely to play a leading role. This retrospective cohort of 250 to 300 cases treated with adjuvant and neoadjuvant will be immunologically characterized using the recommendations of Salgado et al. that a multicentric team of pathologists will take ownership. This evaluation will be counter-appraised.

Once our cohort is immunologically characterized, our project will focus on better understanding the endothelial mechanisms involved: which cells? immunophenotyping of immunity cells. By which vessels? (measurement of densities in blood and lymphatic vessels, density in HEV). By what mechanisms? Do the actors identified in vitro within the Inca project have an in vivo translation

DETAILED DESCRIPTION:
The main objective of this project will be to better understand the behavior of the endothelium in a population of breast cancer where the infiltrate in immune cells is precisely likely to play a leading role. This retrospective cohort of 250 to 300 cases treated with adjuvant and neoadjuvant will be immunologically characterized using the recommendations of Salgado et al., that a multicentric team of pathologists will take ownership. This evaluation will be counter-appraised.

Once our cohort is immunologically characterized, our project will focus on better understanding the endothelial mechanisms involved: which cells? immunophenotyping of immunity cells. By which vessels? (measurement of densities in blood and lymphatic vessels, density in HEV). By what mechanisms? Do the actors identified in vitro within the Inca project have an in vivo translation

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and over
* Confirmed histological diagnosis of breast carcinoma at localized or metastatic stage or colorectal cancer
* Treated at the Oscar Lambret Center or the Henri Becquerel Center between 1/1/2005 and 31/12/2007
* Having undergone surgery for excision of the primary tumor and / or a metastasis
* resected specimen available
* Patients who gave their consent

Exclusion Criteria:

* History of other cancers
* Breast or colic tumors with other histological profiles
* Patient treated for breast or colonic recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with:
  * a breast cancer
  * a colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
correlation between the expression levels of the genes involved in the regulation of endothelial activation and the degree of tumor-infiltrating lymphocytes | 24 months
  The expression of the genes (egfl7, SetD5, other genes and microRNAs) will be evaluated quantitatively by RT-PCR. The amount of RNA obtained corresponds to a relative amount of RNA relative to the amount of RNA measured in a sample used as a reference.
  A semi-quantitative evaluation will also be carried out by in situ hybridization techniques and immunohistochemistry of endothelial expression of endothelial activation regulation markers: 0+ no labeled vessels, 1+ <30% of labeled vessels, 2+ between 30 and 60% of marked vessels, 3+> 60% of marked vessels The lymphocyte infiltration will be evaluated by measuring the ratio between the surface infiltrated by mononuclear cells and the tumor surface (for intratumoral TILS) or stromal (for total stromal TILS). The analysis will be done on H & E slides and the data will be expressed as a percentage.

SECONDARY OUTCOMES:
reproducibility of lymphocyte infiltration assessment on H & E slides | 24 months
study of the subgroups of the cohort with a predominant lymphocytes infiltration cancer | 24 months
  description of subpopulations of immunocompetent cells by specific complementary immunolabeling of CD4 + T lymphocytes (mature T helper lymphocytes expressing the surface protein CD4), cytotoxic CD8 (T lymphocytes expressing the surface protein CD8), T-regulatory (CD25 / FoxP3), B-cell lymphocytes , macrophages and NK (Natural Killer) cells
Cell density description | 24 months
  Description of density in vascular endothelial (CD31 / 34 labeled), lymphatic (LYVE / podoplanin-labeled) and HEV (High endothelial venom MECA79 + (Rat Monoclonal Anti-Peripheral Node Addressin Antibody )) cells and correlation with lymphocyte infiltrate levels
Prognostic value assessment | 24 months
  Evaluate the prognostic value of biomarkers and lymphocytic infiltrate in terms of Global Survival and Survival Without Recurrence
Expression levels of genes involved in the regulation of endothelial activation | 24 months
  In subpopulations of patients treated in neo-adjuvant or metastatic situations: assess the expression levels of genes involved in the regulation of endothelial activation
treatment response data | 24 months
  In subpopulations of patients treated in neo-adjuvant or metastatic situations: assess the treatment response data (chemotherapy in patients with breast cancer, chemotherapy and antiangiogenic in colon cancers)
lymphocytic infiltrate data | 24 months
  For patients treated for breast cancer: study lymphocytic infiltrate data
the existence of a BRCA1 and or BRCA 2 mutation (which are tumour suppressor genes) | 24 months
  For patients treated for breast cancer: assess the existence of a BRCA1 and or BRCA 2 mutation
association between lymphocytic infiltrate data and the RER phenotype (the replication error phenotype) | 24 months
  For patients treated for colon cancer: to study the association between lymphocytic infiltrate data and the RER phenotype
The RER phenotype (the replication error phenotype) | 24 months
  For patients treated for colon cancer: to study the RER phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine Lauridant, MD, Principal Investigator — Centre oscar Lambret de Lille
Locations (2):
- France (2):
  - Centre Oscar Lambret, Lille
  - Centre Henri Becquerel, Rouen